CLINICAL TRIAL: NCT05189093
Title: To Evaluate the Multi-center, Open, Single-arm Phase I/II Clinical Study of Recombinant Humanized Anti-CD47/PD-1 Bifunctional Antibody HX009 Injection in Chinese Patients With Relapsed/Refractory Lymphoma
Brief Title: Recombinant Humanized Anti-CD47/PD-1 Bifunctional Antibody HX009 in Patients With Relapsed/Refractory Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX009-II-02
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phase I dose escalation part,Phase II efficacy exploratory part and the efficacy confirmation part (Experimental): Phase Ib/II efficacy exploration and confirmation phase:
  Four cohorts will be conducted in parallel to initially evaluate the recombinant humanized anti-CD47/PD-1 bifunctional anti HX009 injection.
  The four cohorts in the efficacy exploration phase are:
  Cohort 1: Relapsed/refractory diffuse large B-cell lymphoma; Cohort 2: relapsed/refractory peripheral T-cell lymphoma (except angioimmunoblastic T-cell lymphoma). (except angioimmunoblastic T-cell lymphoma); Cohort 3: relapsed/refractory follicular lymphoma and relapsed/refractory marginal zone lymphoma; Cohort 4: relapsed/refractory EBV-positive non-Hodgkin's lymphoma.
  Interventions: Drug: Recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection

INTERVENTIONS:
Drug: Recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection — There will be a total of 4 cohorts, each cohort will explore 1-2 dose levels, i.e. 10 mg/kg and 15 mg/kg, with an expected enrollment of 40-80 cases. The 10 mg/kg dose level will be enrolled first, the After discussion between the sponsor and the DSC, the 15 mg/kg dose level will be enrolled if necessary. Based on the DMC analysis, the no-trend cohort will be enrolled in a maximum of 10 cases (with the possibility of stopping enrollment halfway through).

SUMMARY:
This study is a multi-center, open, single-arm phase I/II clinical study to evaluate the recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection in Chinese patients with relapsed/refractory lymphoma .

DETAILED DESCRIPTION:
Phase Ib/II efficacy exploration and confirmation phase:

Four cohorts will be conducted in parallel to initially evaluate the recombinant humanized anti-CD47/PD-1 bifunctional anti HX009 injection.

The four cohorts in the efficacy exploration phase are:

Cohort 1: Relapsed/refractory diffuse large B-cell lymphoma; Cohort 2: relapsed/refractory peripheral T-cell lymphoma (except angioimmunoblastic T-cell lymphoma).

(except angioimmunoblastic T-cell lymphoma); Cohort 3: relapsed/refractory follicular lymphoma and relapsed/refractory marginal zone lymphoma; Cohort 4: relapsed/refractory EBV-positive non-Hodgkin's lymphoma. The study will refer to the "Guidelines for Data Monitoring Committees in Drug Clinical Trials (Trial)".

A data monitoring committee will be set up to provide continuous safety monitoring of the study and to provide advice on the dosage and dosing cycle, as well as on the follow-up of the study.

The committee will provide advice on the dosage and cycle of administration, as well as on the decision-making for subsequent extension studies.

Based on the safety data from this study at the 15 mg/kg dose level, during the efficacy exploration phase, the Each cohort will enroll 10-20 subjects, for a total of 4 cohorts, and each cohort will explore 1-2 dose levels, i.e., 10 mg/kg and 15 mg/kg, with an expected enrollment of 40-80 cases. The 10 mg/kg dose level will be enrolled first.

dose level first, and after discussion between the sponsor and the DMC, 15 mg/kg dose level will be enrolled if necessary.

The dose level of 15 mg/kg will be enrolled if necessary after discussion between the sponsor and the DMC. Based on the DMC analysis, the no-trend cohort will be enrolled in a maximum of 10 cases (with the possibility of stop enrollment midway).

The Phase II efficacy confirmation phase will select 1-2 cohorts from the 4 cohorts in the efficacy exploration phase of the study with better safety and efficacy.

1-2 indications with better efficacy to further confirm the efficacy and safety of HX009 injection. Based on the safety and efficacy data from Phase I of this study, the number of cases of subjects in the efficacy confirmation phase will be re-estimated based on statistical principles.

The number of cases of subjects in the validation phase will be re-estimated based on statistical

ELIGIBILITY:
Inclusion criteria：

1. Voluntarily participating in a clinical research study, being fully aware of and informed about the study and signing the Informed Consent Form (ICF).

   Willing to follow and capable of completing all study procedures;
2. Male and Female. Age 18-65 years (including borderline values) in the dose-escalation phase; age 18-70 years (including borderline values) in the efficacy exploration and confirmation phase;
3. lymphoma diagnosed according to the 5th edition of the WHO Classification Criteria for 2022 and meeting the following definition of relapsed or refractory.

   * The Phase Ib efficacy exploration phase will carry out cohort expansion according to the following tumors:

     * Patients with relapsed/refractory diffuse large B-cell lymphoma (including transformed DLBCL): need to have received systemic therapy with at least two standard regimens;
     * Relapsed/refractory peripheral T-cell lymphoma (except angioimmunoblastic T-cell lymphoma): Patients with relapsed/refractory peripheral T-cell lymphoma (except angioimmunoblastic T-cell lymphoma);
     * Relapsed/refractory follicular lymphoma and relapsed/refractory marginal zone lymphoma: at least two standard regimens of systemic therapy are required.
     * Relapsed/refractory EBV-positive non-Hodgkin's lymphoma: at least one systemic regimen is required.
4. an Eastern Cooperative Oncology Group (ECOG) Physical Strength Score of 0 to 2 within 14 days prior to first dose;
5. expected survival ≥ 3 months;
6. good major organ function, i.e., meeting the following criteria:

   * Blood system

     * Absolute neutrophil count (ANC) ≥1.5 × 10/L; with bone marrow invasion, ANC ≥1.0 × 10/L;
     * Platelets ≥75 × 10/L (without bone marrow invasion) and platelets ≥50.0 × 10/L (with bone marrow or spleen invasion);
     * Hemoglobin (HB) ≥90 g/L; HB ≥80 g/L with bone marrow invasion;
   * Liver function

     * Aspartate aminotransferase ≤ 2.0 x ULN, or ≤ 5.0 x ULN for hepatic invasion;
     * Alanine aminotransferase ≤ 2.0 x ULN, or ≤ 5.0 x ULN in hepatic infestation;
     * Total bilirubin ≤ 1.5 × ULN (except in Gilbert's syndrome or with hepatic or pancreatic invasion);
   * Renal function

     * Creatinine clearance ≥ 45 mL/min (calculated according to the Cockcroft-Gault formula, i.e., endogenous creatinine creatinine clearance = [(140 - age) × body weight (kg)]/[0.818 × serum creatinine (umol/L)], for women × 0.85 × calculated result. Sex according to the calculation × 0.85
   * Coagulation

     * International normalized ratio (INR) ≤ 2 times ULN or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
   * Cardiac function

     * Echocardiography: LVEF ≥ 45%.
7. If previous antitumor therapy has been received, the following conditions need to be met:

   * Systemic radiation therapy at intervals of ≥3 weeks from the first dose, localized radiation therapy or bone metastases at Radiation therapy for bone metastasis ≥ 2 weeks;
   * Prior chemotherapy, immunotherapy (CAR-T therapy, etc.), biologic therapy (tumor vaccines, cytokines or cancer-controlling growth factors), targeted therapies, antibody-coupled drugs ≥ 4 weeks or 5 half-lives (whichever is shorter) from the first dose. Previous chemotherapy (CART, etc.), immunotherapy (tumor vaccine, cytokine, or growth factor for cancer control), targeted therapy, antibody-coupled drug ≥ 4 weeks or 5 half-lives from first dose, whichever is shorter;
   * Previous treatment with antitumor Chinese medicine or proprietary Chinese medicine or medicine containing Chinese medicine ingredients for antitumor use and the interval between the first dose is ≥ 1 week;
8. At least one measurable lesion according to Lugano criteria within 4 weeks prior to first dose; measurable Lesions: longest diameter of lymph node >15 mm, invasive lesions elsewhere >10 mm; previously treated lesions with localized therapy such as radiotherapy, if disease progression has been demonstrated and measurable lesions are met. Measurable lesions: longest diameter of lymph node >15 mm, other invasive lesions >10 mm; lesions previously treated with localized therapy, such as radiotherapy, are considered measurable if they have been shown to be progressive and meet the definition of measurable lesions.
9. Female subjects must have a negative serum pregnancy test within 1 week prior to the first dose of study drug; female subjects or male subjects with a partner of childbearing potential agree to use effective contraception (e.g., oral contraceptives, intrauterine devices) for a minimum of 12 months from the time of signing the informed consent form until the last dose of study drug.

Exclusion criteria：

1. Prior history of a malignancy other than skin cancer or carcinoma in situ that is not melanoma (e.g., cervical cancer, bladder cancer, breast cancer, etc.) unless disease-free status has been achieved for 3 years;
2. failure to recover from adverse effects of prior therapy to a CTCAE 5.0 grade score of ≤1, except for residual 3. active gastrointestinal ulcers
3. active peptic ulcer, incomplete intestinal obstruction, active gastrointestinal bleeding and perforation;
4. known history of hereditary or acquired hemolytic or bleeding disorders;
5. subjects with primary or secondary central nervous system (CNS) lymphoma;
6. patients who have received prior targeted therapy with CD47 (including monoclonal antibodies, bispecific antibodies, etc.);
7. patients who have received a blood transfusion or hematopoietic stimulating factor therapy, such as colony-stimulating factor, erythropoietin, erythropoietin, or other stimulating factors within 2 weeks prior to the start of treatment Erythropoietin, thrombopoietin, thrombopoietin, etc;
8. Subjects with an active, or history of, autoimmune disease that is likely to recur or is being treated (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or those at high risk (e.g., who have received organ transplants and need to be treated for immune-suppressant therapy); however, enrollment is permitted in subjects who have :

   * Type 1 diabetes mellitus that has stabilized with the use of fixed-dose insulin;
   * Autoimmune hypothyroidism and adrenal insufficiency requiring only hormone replacement therapy Adenosine insufficiency;
   * Skin diseases that do not require systemic therapy. For example, eczema, a rash that accounts for less than 10% of the body surface, without ophthalmologic symptoms (primarily dry eyes, blepharitis, conjunctivitis, lid adhesions Psoriasis without ophthalmologic symptoms (mainly dry eye, conjunctivitis, lid adhesions, keratitis, and uveitis);
9. major surgery during the Screening Period 28 days prior to the first dose or minor surgery within 2 weeks (except diagnostic surgery), and any elective major surgery during the planned study period;
10. Subjects requiring systemic corticosteroids (dose equivalent to >10 mg prednisone/day) or other immunosuppressive medications within 14 days prior to the first dose or during the study period; the following conditions to >10 mg prednisone/day) or other immunosuppressive medications within 14 days prior to the first dose or during the study period; the following were Enrollment is permitted:

    * Subjects on topical topical or inhaled glucocorticoids;
    * Short-term (≤7 days) use of glucocorticoids for prophylaxis or treatment of non-autoimmune allergic diseases. allergic diseases;
    * Corticosteroids for the replacement therapy of adrenal insufficiency;
    * If high-dose glucocorticoid therapy is urgently needed prior to initiation of study treatment to If high-dose glucocorticoid therapy is urgently needed to control symptoms of lymphoma prior to initiation of study treatment, a tumor evaluation must be completed prior to initiation of treatment.
11. Currently suffers from a serious lung disease requiring treatment or from a previous serious lung disease, interstitial lung disease, interstitial pneumonia. interstitial lung disease, interstitial pneumonia, pulmonary fibrosis, radiation pneumonitis requiring hormone therapy, etc;
12. uncontrolled systemic diseases such as cardiovascular diseases (severe arrhythmia, unstable angina or myocardial infarction within 6 months, etc.) Uncontrolled systemic diseases, such as cardiovascular diseases (severe arrhythmia, unstable angina or myocardial infarction within 6 months), diabetes mellitus, hypertension, etc. 13;
13. arterial or venous thrombosis or embolic events within 3 months prior to the first dose, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis or pulmonary embolism;
14. being positive for human immunodeficiency virus or having other acquired, congenital immunodeficiency diseases. History of organ transplantation or allogeneic stem cell transplantation;
15. active tuberculosis disease or latent tuberculosis infection;
16. Subjects with active hepatitis B or hepatitis C. Hepatitis B patients: HBsAg or HBcAg positive. Except for the following:

    * If HBcAg positive, not associated with HBsAg positivity, negative DNA test (<20 IU or lower limit of local laboratory normal) and subject to periodic DNA testing during the study period;
    * Cured Hepatitis C subjects (negative HCV RNA test);
17. subjects with severe active infection within 2 weeks prior to the first dose of study drug;
18. subjects with a known history of severe allergic reactions to large protein preparations or to any of the components of the test drug (CTC); or 18. a known subject with a previous severe allergic reaction (CTCAE 5.0 ≥ 3) to a large protein preparation or to any of the components of the test drug;
19. participation in a clinical trial of another drug within 4 weeks prior to the first dose;
20. alcohol dependence or a history of drug or substance abuse within the last 1 year
21. previous history of definite neurological or psychiatric disorders, such as epilepsy, dementia, poor adherence;
22. women who are pregnant or breastfeeding;
23. Subjects who have received any live or attenuated vaccine within 28 days prior to the first dose of study drug. If enrolled, subjects must not receive any live or attenuated vaccine during the study period or within 180 days of the last dose of HX009. Live Vaccines. Subjects vaccinated with inactivated, mRNA, viral vector, and labeled protein COVID-19 vaccines are eligible to participate in the study. Subjects vaccinated with inactivated, mRNA, viral vector and labeled protein COVID-19 vaccines are eligible to participate in the study and the vaccination timeline should follow local guidelines;
24. subjects who, in the opinion of the Investigator, are otherwise unsuitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) of patients with solid tumors treated with HX009 per Investigator Assessment | Tumor assessment every 6 weeks (±7 days)，up to 1 year
  Objective response rate (ORR) assessed according to the evaluation criteria of each tumor type

SECONDARY OUTCOMES:
6 months and 12 months progression-free survival (PFS ) | Approximately 1 year
  PFS is defined as the time from the start of the first dose and the first documented disease progression using RECIST 1.1 criteria or death of any cause.
Complete Remission Rate (CRR) | Approximately 1 year
  Disappearance of all target lesions, no new lesions appearing
Duration of Remission (DOR) | Tumor assessment every 6 weeks (±7 days),up to 1year
  The DOR is defined as the time from the first recorded response (CR or PR) to the first recorded tumor progression or death due to any cause.
Disease Control Rate (DCR) | Tumor assessment every 6 weeks (±7 days),up to 1 year
  The DCR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response, or Partial Response, or Stable Disease using RECIST 1.1 criteria.
Incidence and severity of AE and SAE, laboratory tests and vital signs（Including ：heart rate, blood pressure, respiration,temperature.）; | All AEs up to 28 days after the last dose of study drug,Or other tumor treatment programs have been started (the earlier date shall prevail); irAE should be followed up to 90 days after the last dose, or other tumor treatment programs have been started
  Adverse events (AEs) determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: Tmax | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: Tmin | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: Cmin | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: Cavg | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: AUCss | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: t1/2 | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: λz | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: CLss/F | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: Vz/F | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: DF | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: AUC0-t | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: AUC0-∞ | Approximately 1 year
  Key pharmacokinetic parameter
Pharmacokinetic parameters of recombinant humanized anti-CD47/PD-1 bifunctional antibody HX009 injection: AUCext% | Approximately 1 year
  Key pharmacokinetic parameter
Peak plasma concentration (Cmax) of HX009 in patients with relapsed/refractory lymphoma | Approximately 1 year
  Key pharmacokinetic parameter
Antidrug antibodies (ADA) | Approximately 1 year
  Key pharmacokinetic parameter
Neutralizing antibodies (Nab) after treatment (ADA-positive individuals only) | Approximately 1 year
  Key pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciense, Beijing, Beijing Municipality, China